CLINICAL TRIAL: NCT01042210
Title: Genotype-phenotype Associations of Agouti-related Peptide (AgRP) in Postpartum Period in Preeclamptic and Non-preeclamptic Women and Their Offspring
Brief Title: Agouti-related Peptide (AgRP) in Healthy Mothers and Mothers With Preeclampsia and Their Offspring
Status: Completed | Type: Observational
Sponsor: Masaryk University (Other)
Responsible Party: prof. MUDr. Anna Vašků, CSc., Head of the department of pathological physiology, Department of pathological physiology, Faculty of Medicine, Masaryk university, Brno
Other Study IDs: MU-JBV-PPM1
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Last update posted 2010-01-05 (Estimated); Status verified 2009-11

CONDITIONS: Preeclampsia
Keywords: preeclampsia; agouti-related peptide; intrauterine growth; birth weight; Intrauterine growth restriction due to preeclampsia
MeSH Terms: conditions — Pre-Eclampsia; Birth Weight

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood, umbilical blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Mothers, preeclampsia: Mothers with preeclampsia diagnosed according to the Guidelines by the Czech Society of obstetrics and gynecology as development of hypertension after the 20th week of pregnancy (systolic blood pressure, ≥140 mmHg; and/or diastolic blood pressure, ≥90 mmHg; measured at rest on two consecutive occasions at least 24 h apart) in previously normotensive women, and the onset of proteinuria (>300 mg of urinary protein/L over 24 h).
- Newborns, physiological pregnancy-delivery: The newborns from the physiological pregnancies with spontaneous, uncomplicated delivery.
- Newborns, pregnancy with preeclampsia: Newborns from the pregnancies complicated by preeclampsia.
- Mothers, Physiological pregnancy-labour: The cohort of non-preeclamptic mothers with physiological, uncomplicated conception, pregnancy and delivery.

SUMMARY:
The study is focused on the investigation of possible associations between plasma/serum levels of agouti related peptide (AgRP) and its genetic background in healthy women with physiological pregnancy (non-preeclamptic) and women with preeclampsia, in the postpartum period, and in their offspring.

DETAILED DESCRIPTION:
The study is focused on investigation of possible genotype-phenotype interactions of agouti-related peptide (AgRP) in postpartum non-preeclamptic women and preeclamptic women and in their offspring.

ELIGIBILITY:
Inclusion Criteria:

* For preeclampsia:

  * development of hypertension after the 20th week of pregnancy (systolic blood pressure, ≥140 mmHg; and/or diastolic blood pressure, ≥90 mmHg; measured at rest on two consecutive occasions at least 24 h apart) in previously normotensive women, and the onset of proteinuria (>300 mg of urinary protein/L over 24 h)
  * single-fetus pregnancy
  * age range 18-35 y
  * no preconceptional history of hypertension
* For mother with physiological pregnancies:

  * uncomplicated
  * spontaneous conception
  * single-fetus pregnancy
  * age range 18-35 y
  * spontaneous uncomplicated delivery
  * no history of preconceptional hypertension

Exclusion Criteria:

* For preeclampsia:

  * multiple pregnancy
  * preeclampsia superimposed to chronic hypertension preceding pregnancy
  * kidney disease
  * fetal malformations
* For mothers with physiological pregnancies:

  * in vitro fertilization
  * fetal malformations
  * multiple pregnancy
  * events of bleeding

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients of the Masaryk university afilliated hospital, Clinic of Obstetrics and Gynecology,hospitalized due to preeclampsia or healthy women with uncomplicated conception, pregnancy and delivery that came to give birth at the Clinic. Along with the mothers, their offspring in included in the study. The study population originated from a static region of the Czech Republic - South Moravia.
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2005-01; Primary Completion 2006-03 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
plasma/serum level of agouti/related peptide in peripheral blood in postpartum mother | 2-4 hours postpartum
Plasma level of agouti-related peptide in umbilical cord blood from the newborn | immediately postpartum

SECONDARY OUTCOMES:
maternal weight gain during pregnancy | using postpartum and peripartum data
birth weight of the newborn | immediately postpartum
maternal preconceptional BMI | anamnestic information

CONTACTS AND LOCATIONS:
Overall Officials: Julie Bienertova-Vasku, MD.,, Ph.D., Principal Investigator — Department of Pathological Physiology, Faculty of Medicine, Masaryk University; Anna Vasku, prof. Ph.D., Study Director — Department of Pathological Physiology, Faculty of Medicine, Masaryk University; Petr Bienert, Dr., Study Director — Department of Pathological Physiology, Faculty of Medicine, Masaryk University
Locations (1):
- Masaryk university affiliated hospital, Clinic of Obstetrics and Gynecology, Brno, Moravia, Czechia

REFERENCES:
- [Background] Wagner CG, McMahon CD, Marks DL, Daniel JA, Steele B, Sartin JL. A role for agouti-related protein in appetite regulation in a species with continuous nutrient delivery. Neuroendocrinology. 2004;80(4):210-8. doi: 10.1159/000082735. Epub 2004 Dec 13. PMID 15604600
- [Background] Tamura H, Kamegai J, Shimizu T, Ishii S, Sugihara H, Oikawa S. The effect of agouti-related protein on growth hormone secretion in adult male rats. Regul Pept. 2005 Feb 15;125(1-3):145-9. doi: 10.1016/j.regpep.2004.08.012. PMID 15582725
- [Background] Gavrila A, Chan JL, Miller LC, Heist K, Yiannakouris N, Mantzoros CS. Circulating melanin-concentrating hormone, agouti-related protein, and alpha-melanocyte-stimulating hormone levels in relation to body composition: alterations in response to food deprivation and recombinant human leptin administration. J Clin Endocrinol Metab. 2005 Feb;90(2):1047-54. doi: 10.1210/jc.2004-1124. Epub 2004 Nov 16. PMID 15546902
- [Background] Hoggard N, Johnstone AM, Faber P, Gibney ER, Elia M, Lobley G, Rayner V, Horgan G, Hunter L, Bashir S, Stubbs RJ. Plasma concentrations of alpha-MSH, AgRP and leptin in lean and obese men and their relationship to differing states of energy balance perturbation. Clin Endocrinol (Oxf). 2004 Jul;61(1):31-9. doi: 10.1111/j.1365-2265.2004.02056.x. PMID 15212642